CLINICAL TRIAL: NCT05414071
Title: The Impact of a Digital Artificial Intelligence System on the Monitoring and Self-management of Non-motor Symptoms in People With Parkinson's
Brief Title: Clinical Investigation of NMS Assist
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study sponsor has changed and is no longer the University of Plymouth. A new record is being created under the updated sponsor.
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Associate Professor of eHealth, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AM1000398
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson
Keywords: Parkinson Disease; Self-Management; Telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NMS Assist (Experimental): NMS Assist provides a system of linking PwP, CPs, and healthcare providers (HCPs) to monitor and empower self-management of non-motor symptoms through the use of a mobile app and web portal.
  Interventions: Device: NMS Assist

INTERVENTIONS:
Device: NMS Assist — The system enables people with Parkinson's and their care partners to complete questionnaires about symptoms and burden and share that information with their care team. They can also access self-help resources and materials about managing non-motor symptoms. Healthcare providers have a dashboard that flags any worsening symptoms or discrepancies between PwP and CP reports, enabling their to prioritise care and quickly see the status of their patients. The system also enables PwP or CPs to request healthcare contact.

SUMMARY:
Parkinson's can cause a wide range of non-motor symptoms (NMS), including pain and problems with mental health, memory and sleep. These affect the quality of life of people with Parkinson's (PwP) and their care partners (CP). If these issues are not recognised and managed quickly, they can result in escalating problems. Many PwP are unsure of the extent and variety of the NMS and how simple adjustments at home could improve them. We have developed a digital system, NMS Assist, to help PwP monitor their non-motor symptoms and develop skills to self-manage them.

Such a tool needs to be simple to use, safe and effective. We will ask 60 PwP, CP and members of their Parkinson's healthcare team to use NMS Assist for 12 months, and we will monitor how they use the tool. PwP and CPs will be asked if they feel more knowledgeable and confident to manage their own symptoms whilst being better able to discuss a problem with their healthcare professional.

A smaller group of the participants will discuss their experiences in more detail to help pinpoint aspects that work well and those needing adjustment and development. Members of the healthcare team will be asked to assess any improvement in communication with PwP and CPs.

It is thought that the use of this system will result in improved quality of life and increased knowledge and confidence for managing symptoms while safely reducing the time spent by health care professionals on manageable non-motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and comply with intervention requirements
* 18 years or older
* Be fluent in English
* Not resident in a care or nursing home
* Ambulant
* Have compatible smartphone/data access
* Normally under the care of the Parkinson's service in the participating organisation
* Participant's HCP in the participating organisation consented to participate in the study

Exclusion Criteria:

* Secondary cause of parkinsonism
* Significant cognitive impairment or a diagnosis of Parkinson's disease dementia
* Living in residential care facilities
* Previous involvement in development or testing of the NMS Assist system
* Significant comorbidity, which in the opinion of the chief investigator would preclude safe participation in the study or protocol compliance (e.g. life expectancy <6 months)
* In a dependent/unequal relationship with anyone involved in the research or care teams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient (and care partner) activation | Assessed monthly for 12 months
  Patient Activation Measure (and caregiver version) will be used to evaluate their confidence, knowledge, and skills at non-motor symptom self-management

SECONDARY OUTCOMES:
Presence of non-motor symptoms | Measured at patients' discretion throughout intervention (12 months)
  Measured using the Non-Motor Symptoms Questionnaire (NMSQ), patients tick 'yes' or 'no' for each symptom listed
Frequency and severity of non-motor symptoms | Measured at baseline, 6, and 12 months
  Measured using the Movement Disorder Society Non-Motor Symptoms Scale (MDS-NMS), where higher scores indicate greater frequency and/or severity
Short-form self-assessment of functioning and well-being related to Parkinson's disease | Measured at patients' discretion throughout intervention (12 months)
  Measured using the short-form Parkinson's Disease Questionnaire (PDQ-8), patients indicate the frequency with which they experience certain issues
Long-form self-assessment of functioning and well-being related to Parkinson's disease | Measured at baseline, 6, and 12 months
  Measured using the long-form Parkinson's Disease Questionnaire PDQ-39, patients indicate the frequency with which they experience certain issues
Carer well-being and quality of life | Measured at care partners' discretion throughout intervention (12 months)
  Measured using the Parkinson Disease Questionnaire for care partners; care partners indicate the frequency with which they experience certain issues
Health status | Measured at baseline, 6, and 12 months
  Measured using the EQ-5D-5L; higher scores on the EQ-5D-5L descriptive system indicate worse health problems in the specific dimension whereas a high score in the EQ VAS indicates better health on the day of the questionnaire
Mental well-being | Measured at baseline, 6, and 12 months
  Measured using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS); Scores range from 14 to 70 (on the 14 item version) and higher scores indicate greater positive mental wellbeing
Adverse events | Throughout 12 months
  Adverse Event Reporting
Clinical safety | Throughout 12 months
  Record of any events missed
Healthcare contacts | Throughout 12 months
  Number of PwP-initiated contacts with healthcare team (through the 'request healthcare contact' feature) and the number of HCP-initiated contacts (due to system flagging PwP based on PwP and CP-reported outcomes), recorded by the system
Technical and implementation issues | Throughout 12 months
  Technical issues identified from the system use data and by participants and process measures relating to service delivery
Quantitative usability | 6 and 12 months
  System Usability Scale, out of 100 with higher scores indicating better usability
Acceptability | 3, 6, and 12 months
  Acceptability and usability feedback from semi-structured interviews
System use and compliance | Throughout 12 months
  Data collected via the system about users engagement with the system (e.g. number of times accessed, length of time accessed, features used)
Engagement | 3, 6, and 12 months
  Qualitative feedback from participants
Costs | Throughout 12 months
  Cost analysis will be used to examine the factors impacting costs for implementing the system

IPD SHARING:
Plan to Share IPD: Undecided
Data belongs to the study sponsor (the University of Plymouth) and deidentified data will be made available in line with the data sharing policy developed with Parkinson's UK and PPI representatives.

REFERENCES:
- [Derived] Meinert E, Milne-Ives M, Chaudhuri KR, Harding T, Whipps J, Whipps S, Carroll C. The Impact of a Digital Artificial Intelligence System on the Monitoring and Self-management of Nonmotor Symptoms in People With Parkinson Disease: Proposal for a Phase 1 Implementation Study. JMIR Res Protoc. 2022 Sep 26;11(9):e40317. doi: 10.2196/40317. PMID 36155396